CLINICAL TRIAL: NCT05062005
Title: Induction Chemotherapy+Chemoradiotherapy vs. Chemoradiotherapy for Locally Advanced Nasopharyngeal Carcinoma
Brief Title: ICCRT vs. CRT for Locally Advanced Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Chen Yong, Professor, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCICCRTvCRT
Record Dates: First submitted 2021-09-07; First posted 2021-09-30 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Locally Advanced Nasopharyngeal Carcinoma
MeSH Terms: interventions — Induction Chemotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Induction Chemotherapy+Chemoradiotherapy (Other)
  Interventions: Drug: Induction Chemotherapy; Drug: Concurrent Chemotherapy; Radiation: Definitive Radiotherapy
- Chemoradiotherapy (Other)
  Interventions: Drug: Concurrent Chemotherapy; Radiation: Definitive Radiotherapy

INTERVENTIONS:
Drug: Induction Chemotherapy — Induction regimens: TP (docetaxel 75 mg/m²; cisplatin 75 mg/m²) Q3w, TPF (docetaxel 60 mg/m²; cisplatin 60 mg/m²; 5-fluorouracil 600-750 mg/m² per day, continuous intravenous infusion d1-5) Q3w, or GP (gemcitabine: 1000 mg/m2 d1, d8; cisplatin 80 mg/m2) Q3w.
  Arms: Induction Chemotherapy+Chemoradiotherapy
Drug: Concurrent Chemotherapy — Cisplatin 100 mg/m², Q3w.
Radiation: Definitive Radiotherapy — For all patients, the prescribed dose is 66-70 Gy (once a day, 5 times a week).

SUMMARY:
This trial is a multi-center phase III clinical trial. The purpose of this trial is to explore whether concurrent chemoradiotherapy is not inferior to induction chemotherapy combined with concurrent chemoradiotherapy in patients with locally advanced nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years old;
2. Pathologically confirmed non-keratinizing nasopharyngeal carcinoma;
3. Stage T3-4N0-1 (according to the UICC/AJCC 8th);
4. No distant metastasis;
5. Have not received anti-cancer treatment in the past;
6. ECOG (Eastern Cooperative Oncology Group of the United States): 0-1;
7. Adequate hematologic, hepatic and renal function.

Exclusion Criteria:

1. The purpose of treatment is palliative;
2. Diagnosed with other malignant tumors at the same time;
3. Malignant tumor history;
4. Pregnancy or breastfeeding, or expect to become pregnant during the clinical trial period;
5. Combined serious illness.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 447 (Estimated)
Dates: Start 2021-09-22 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
FFS (Failure-free Survival) | 3 year
  Defined as the time from randomization to tumor recurrence, distant metastasis, or death due to any reason, whichever occurs first. Patients who withdraw or who are lost to follow-up will be censored at the date last known to be alive and progression free. Patients not having an event will be censored at the date last seen alive.

SECONDARY OUTCOMES:
OS (Overall Survival) | 3 year
  Defined as the time from randomization until death from any cause. Patients who withdraw or who are lost to follow-up will be censored at the date last known to be alive. Patients remaining alive throughout the duration of the study will have their survival time censored on the date last seen alive.
LRFS (Locoregional Recurrence-free Survival) | 3 year
  Defined as the time from randomization to local or regional recurrence. Patients who withdraw or who are lost to follow-up will be censored at the date last known to be alive and recurrence free. Patients not having an event will be censored at the date last seen alive.
DMFS (Distant Metastasis-free Survival) | 3 year
  Defined as the time of randomization to the appearance of distant metastasis. Patients who withdraw or who are lost to follow-up will be censored at the date last known to be alive and metastasis free. Patients not having an event will be censored at the date last seen alive.
AE (Adverse events) | 3 year
  Adverse events during the treatment period will be assessed according to the Common Terminology Criteria for Adverse Events (CTCAE, version 5.0). Late AE of radiotherapy will be assessed according to RTOG criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No